CLINICAL TRIAL: NCT00721981
Title: A Non-interventional Study for Evaluation of the Clinical Treatment and Patient Values and Preferences of Patients Suffering From Advanced Non-small Cell Lung Cancer (NSCLC) Undergoing Chemotherapy. With Special Focus on Patients Who Are in Transition From First Line to Second Line Treatment
Brief Title: An Evaluation of the Clinical Treatment and Patient Values and Preferences of Patients Suffering From Advanced Non-small Cell Lung Cancer (NSCLC) Undergoing Chemotherapy
Status: Terminated | Type: Observational
Why Stopped: Low Recruitment
Sponsor: AstraZeneca (Industry)
Responsible Party: Chris Teale, Director Global Pricing & Market Access (Oncology), AstraZeneca UK Limited
Other Study IDs: NIS-ODE-DUM-2008/1
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: patient preference; oncology; chemotherapy; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Patient Preference; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Regular treatment for non-small cell lung cancer (NSCLC)

SUMMARY:
The main purpose of this study is the identification, description, and segmentation of non-small cell lung cancer (NSCLC) patients based on their value appraisal of treatment outcomes and all intermediate states of health, to obtain patient preferences in direct correlation with clinical data from patients suffering from NSCLC (stage IIIB / IV) who are in transition from 1st to 2nd line treatment, and to gain utility scores by health state derived from patients' perceived value and taken from their perspective.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from non-small cell lung cancer (NSCLC) with clinical stage IIIB and IV tumours
* Patients with one chemotherapy regimen (first line treatment) (adjuvant chemotherapy following surgery is also regarded as first line treatment)
* Patients who are in transition from first to second line treatment
* Patients who signed an informed consent

Exclusion Criteria:

* Chemotherapy naïve patients
* Patients ever enrolled in clinical studies treating non-small cell lung cancer (NSCLC) with chemotherapy (during 1st and 2nd line chemotherapy)
* Patients who ever had chemotherapy for an indication other than NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from non-small cell lung cancer (NSCLC) (stage IIIb and IV) undergoing chemotherapy, who are in transition from 1st to 2nd line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-04; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To obtain patient preferences in direct correlation with clinical data from patients suffering from NSCLC stage IIb/IV who are in transition from 1st line to 2nd line treatment | once only, 4-6 weeks after switch from 1st to 2nd line chemotherapy

SECONDARY OUTCOMES:
current medical practice treatment objectives and modalities side effects | once only, 4-6 weeks after switch from 1st to 2nd line chemotherapy
socioeconomic status and demographics patients' perception of their health status and treatment patient values and patient preferences | once only, 4-6 weeks after switch from 1st to 2nd line chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Teale, Study Director — AstraZeneca UK Limited, Alderley House, Alderley Park, Macclesfield SK10 4TF, Cheshire, United Kingdom, Phone: +44 1625 516549 Fax: +44 1625 518982; Oliver Fietz, PhD, Study Chair — AstraZeneca GmbH, Tinsdaler Weg 18322880, Wedel, Germany, Phone: +49 (0) 4103 708-3096 Fax: +49 (0) 4103 708-7-3096; Helge Bischoff, MD, Principal Investigator — Thoraxklinik Heidelberg, gGmbH, Amalienstr. 5, 69126 Heidelberg, Germany, Phone: +49 (0) 6221 396-1304 Fax: +49 (0) 6221 396-1305
Locations (8):
- Germany (8):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Heidelberg
  - Research Site, Hemer
  - Research Site, Karlsruhe
  - Research Site, Löwenstein
  - Research Site, München
  - Research Site, Trier